CLINICAL TRIAL: NCT02292888
Title: Can Changes in LVOT VTI Before and After Passive Leg Raising (PLR) Test Serve as a Sensitive Indicator for Changes in SV and CO and Hence Volume Responsiveness ?
Brief Title: Can Changes in Velocity Time Integral Serve as a Sensitive Indicator for Monitoring Changes in Stroke Volume ?
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fortis Hospital, India (Other)
Responsible Party: Principal Investigator, Saikat Bandyopadhyay, MD, Consultant Cardiac Anesthesiologist & Intensivist, Fortis Hospital, India
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Screening
Other Study IDs: FortisH
Record Dates: First submitted 2014-11-13; First posted 2014-11-17 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Ischemic Heart Disease
Keywords: Doppler VTI TEE SV volume responsiveness
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- patients with LVEF >40% (Active Comparator): Correlation between hemodynamic variable : SV and echocardiographic variable : Doppler VTI will be compared before and after Passive Leg Raising (PLR) test.
  Interventions: Other: Passive Leg Raising (PLR) test
- patients with LVEF < or equal to 40% (Active Comparator): Correlation between hemodynamic variable : SV and echocardiographic variable : Doppler VTI will be compared before and after Passive Leg Raising (PLR) test.
  Interventions: Other: Passive Leg Raising (PLR) test

INTERVENTIONS:
Other: Passive Leg Raising (PLR) test — Passive Leg Raising (PLR) test

SUMMARY:
Hypothesis: A validated technique to measure cardiac output (CO) using echocardiography is to calculate stroke volume from the product of LVOT area and LVOT VTI and multiplying the product with heart rate ( CO = SV x H/R; SV = LVOT area x LVOT VTI ).

The LVOT diameter for an individual is more or less a constant measurement. Therefore using the formula mentioned above (SV = LVOT area x LVOT VTI), if the LVOT area is constant, then SV should be proportional to the VTI. This means if a PLR manoeuvre or fluid bolus helps to achieve a rise in SV, then it should be reflected in an increase in VTI as well. If this assumption is true, then an increase in the value of VTI from baseline after fluid challenge (10-15%), should identify a volume responsive patient.

DETAILED DESCRIPTION:
Can changes in LVOT VTI before and after passive leg raising (PLR) test serve as a sensitive indicator for changes in SV and CO and hence volume responsiveness ?

What is Doppler LVOT VTI? Placing a Pulsed Wave Doppler gate on the LVOT immediately below the opening of the aortic valve while aligning the Doppler beam as parallel to the LVOT/aortic axis as possible with an angle of Doppler alignment <20˚, one may obtain Doppler flow velocity measurements which can help measure the LVOT VTI (Velocity Time Integral). If one integrates this velocity profile between two time points (i.e., calculates the area under the curve), the distance traversed of "a region of blood" flowing during this period may be estimated. Since flow velocity is not constant throughout a flow cycle, all of the flow velocities during the entire ejection period is integrated to measure "distance traversed" of this "region of blood." This integration of flow velocities in a given period of time is called the velocity-time integral (VTI)(1) and yields length or distance (measured in cm).

Goal: Whether VTI (LVOT) measured from the deep transgastric (deep TG) or transgastric long axis (TG LAX ) views reflect changes in stroke volume(SV) and hence cardiac output (CO) measured by the gold standard method (PA CCO by thermodilution) before and after passive leg raising test (PLR).

Hypothesis: A validated technique to measure cardiac output (CO) using echocardiography is to calculate stroke volume from the product of LVOT area and LVOT VTI and multiplying the product with heart rate ( CO = SV x H/R; SV = LVOT area x LVOT VTI ).

The LVOT diameter for an individual is more or less a constant measurement. Therefore using the formula mentioned above (SV = LVOT area x LVOT VTI), if the LVOT area is constant, then SV should be proportional to the VTI. This means if a PLR manoeuvre or fluid bolus helps to achieve a rise in SV, then it should be reflected in an increase in VTI as well. If this assumption is true, then an increase in the value of VTI from baseline after fluid challenge (10-15%), should identify a volume responsive patient.

Why do the investigators wish to do the study? A significant improvement in the field of anesthesiology would occur if we could have a simple yet accurate relatively non-invasive tool to correctly assess fluid responsiveness. Excessive fluid infused in the operating room would prolong mechanical ventilation and stay in the ICU and negatively affect the prognosis of the patient. While monitoring with CCO PA catheter considerable adds to the expense, it has its own complications and as may not be indicated in majority of operative cases. A simple non invasive tool using TEE can significantly add to our understanding of hemodynamics and help guide fluid therapy. If our assumption proves to be correct, then it could be a simple, yet rapid bedside indicator of CO. It could be used as a simple tool to assess fluid responsiveness.

The fundamental reason why a fluid challenge (PLR or fluid boluses) is used is to assess whether there is an increase stroke volume in response to it (2). If the fluid loading fails to improve the stroke volume the fluid challenge/loading serves no useful purpose. In normal physiological conditions both the ventricles operate on the ascending limb of the Frank-Starling curve. Once the left ventricle starts functioning on the 'flat' portion of the Frank-Starling curve, fluid loading has little or no effect on stroke volume. If LVOT VTI could be shown to reflect SV adequately then it will be a relatively simple non invasive dynamic bedside tool to test if fluid boluses are resulting in an increase in VTI hence the SV.

Volume responsiveness has been assessed in literature by measuring the response to fluid boluses or to PLR. Thus a positive test where after a PLR, VTI increased significantly reflecting a positive change in SV and CO, more fluid would be required. Whereas if during PLR, CO and SV diminished reflected by a decrease in the VTI value compared to baseline, the subject would be unlikely to respond to fluid therapy and probably would require inotropic support.

Why PLR ? A recent meta-analysis (3), which pooled the results of eight recent studies, confirmed the excellent value of PLR to predict fluid responsiveness in critically ill patients with a global area under the receiver operating characteristic curve of 0.95.

Limitations of using Doppler VTI: However, use of these equations entails a number of assumptions, including (a) laminar blood flow in the area interrogated, (b) a flat or blunt flow velocity profile such that the flow across the entire CSA interrogated is relatively uniform, and (c) Doppler angle of incidence between the Doppler beam and the main direction of blood flow is less than 20 degrees, so that the underestimation of the flow velocity is less than 6%.

Study population: 50 adult patients undergoing coronary artery bypass surgery. Materials & Methods: After institutional ethics committee approval and personal informed consent, 50 patients undergoing elective coronary artery bypass surgery would be included into the study. Patients with significant arrhythmias, concomitant aortic aneurysms, and esophageal pathology precluding the use of TEE would be considered ineligible for the study.

Patients would be divided into two groups. Patients with normal LV function or mild LV systolic dysfunction (LVEF >40%)(4), assessed by preoperative echocardiography would comprise Group 1, whereas those with preoperative LV moderate to severe systolic dysfunction (LVEF <40%)(4) would be designated to Group 2.

Anesthetic protocol: Patients would be fasted for 8 hours preceding the operation. No i.v. fluids would be administered during this period. Patients would be pre-medicated with their usual cardiovascular medication and 1mg of Lorazepam the night before and would receive 1-2 mg of Midazolam at arrival to the operation theatre. After initiating standard monitoring (ECG, Pulse oximetry, NBP) invasive lines would be introduced under local anesthetic infiltration while the patient would receive supplemental oxygen via facemask. Induction of anesthesia would include 0.05 mg kg_1 Midazolam and 5 mcg kg_1 Fentanyl in addition to Sevoflurane 3-5% titrated to loss of eyelash reflex. Tracheal intubation would be facilitated by Rocuronium 0.1 mg kg_1. Anaesthesia would be maintained by Sevoflurane 1.5-2% titrated to an end tidal value of >1.5%and above supplemented by additional doses of fentanyl up to a total dose of 15-20 mg kg_1. All patients would receive 500 ml of lactated Ringer solution during the induction period.

Hemodynamic and Echocardiographic monitoring. A 7.0Fr triple lumen central line, a 8.5 Fr PA sheath and 7.0 Fr CCO (Continuous Cardiac Output) PA catheter and a 16 G femoral arterial canula would be introduced prior to induction of anesthesia under light sedation and local anesthesia. ''''A Philips HD 11XE ultrasound machine (Andover, USA) and transesophageal multiplane echocardiographic probe would be used in all patients. After a comprehensive TEE examination the probe would be positioned to record images from either a deep TG or TGLAX views. Images would be recorded for off-line evaluation. A Board certified echocardiographer proficient in TEE would perform all echocardiographic measurements. Offline echocardiographic measurements would be done by a trained echocardiographer who would be blinded to the study protocol. All hemodynamic measurements will be recorded by a dedicated research nurse.

Experimental protocol: After the induction of anesthesia and initiation of hemodynamic monitoring the patients would be stabilized as necessary and observed for 10-15 min. No further interventions would be allowed during this period, including further fluid administration, changes in anesthetic concentrations or manipulations with inotropic or vasoconstrictor concentrations. A period of at least 5 min of stable BP, heart rate, CVP, and continuous cardiac output would be required before obtaining the baseline set of hemodynamic measurements. A passive leg raising (PLR) maneuver (45%) using protocol described before* in literature would be performed and changes in hemodynamic and echocardiographic parameters would be measured within 1 minute post PLR. The same sequence of PLR and echocardiographic and hemodynamic measurements would be repeated after the end of the operation and before the transfer to the ICU. No measurements would be carried out in the presence of hemodynamic instability or immediately following changes of inotropic or anesthetic medications.

The first set of measurements (HR, MAP, VTI, SV, CO, LVEF and LVOT area ) would be obtained in the semi-recumbent position (45°; designated 'baseline'). Then, the lower limbs would be lifted while straight (45°) with the trunk lowered in the supine position. The second set of measurements of (designated 'during PLR') was obtained during leg elevation, at the moment when VTI plateaued at its highest value. The stroke volume with CCO monitor would be recorded at the moment when it plateaued at its highest value.

NB. Why record changes in VTI/SV etc . within 1 minute post PLR ? Because the maximal hemodynamic effects of PLR occur within the first minute of leg elevation, it is important to assess these effects with a method that is able to track changes in cardiac output or stroke volume on a real-time basis.(5)

NB. Passive leg raising. The passive leg raising test consists in measuring the hemodynamic effects of a leg elevation up to 45°. A simple way to perform the postural maneuver is to transfer the patient from the semirecumbent posture to the passive leg raising position by using the automatic motion of the bed.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing CABG (coronary artery bypass surgery )

Exclusion Criteria:

* Significant arrhythmias
* Concomitant aortic aneurysms,
* Esophageal pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-12; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Whether a change in Doppler VTI before and after passive leg raising test (PLR) correctly reflects changes in stroke volume measured by CCO PA catheter | within 1 minute
  the 3 highest values of VTI post PLR measured between 30 seconds to maximum of 60 seconds post PLR test are to be used and their mean value is to be compared with the mean stroke volume (SV) recorded by the CCO monitor during the same period.

REFERENCES:
- [Background] 1. Reich DL Gregory W. Perioperative Transesophageal Echocardiography: A Companion to Kaplan's Cardiac Anesthesia by . Fischer 1st edition. Chapter 4.
- [Result] Marik PE, Monnet X, Teboul JL. Hemodynamic parameters to guide fluid therapy. Ann Intensive Care. 2011 Mar 21;1(1):1. doi: 10.1186/2110-5820-1-1. PMID 21906322
- [Result] Cavallaro F, Sandroni C, Marano C, La Torre G, Mannocci A, De Waure C, Bello G, Maviglia R, Antonelli M. Diagnostic accuracy of passive leg raising for prediction of fluid responsiveness in adults: systematic review and meta-analysis of clinical studies. Intensive Care Med. 2010 Sep;36(9):1475-83. doi: 10.1007/s00134-010-1929-y. Epub 2010 May 26. PMID 20502865
- [Result] Atherton JJ. Screening for left ventricular systolic dysfunction: is imaging a solution? JACC Cardiovasc Imaging. 2010 Apr;3(4):421-8. doi: 10.1016/j.jcmg.2009.11.014. PMID 20394904
- [Result] Monnet X, Rienzo M, Osman D, Anguel N, Richard C, Pinsky MR, Teboul JL. Passive leg raising predicts fluid responsiveness in the critically ill. Crit Care Med. 2006 May;34(5):1402-7. doi: 10.1097/01.CCM.0000215453.11735.06. PMID 16540963